CLINICAL TRIAL: NCT06713967
Title: Comparison of Outcome of Pregnant Females with Polycystic Ovarian Syndrome with or Without Glucophage
Brief Title: Comparison of Pregnancy Outcomes in Women with Polycystic Ovarian Syndrome with and Without Glucophage
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Health Sciences Lahore (Other)
Responsible Party: Principal Investigator, Dr. Amina Waheed, Post Graduate Resident, University of Health Sciences Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Exp126
Record Dates: First submitted 2024-11-26; First posted 2024-12-03 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Polycystic Ovarian Syndrome (PCOS); Pregnancy Outcomes
MeSH Terms: conditions — Polycystic Ovary Syndrome | interventions — Metformin; Standard of Care; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Glucophage Treatment Group (Experimental): In this arm, participants will receive a standard diet and exercise plan along with Glucophage (metformin). Metformin will be administered starting at 500 mg daily and gradually increased to 1500 mg daily for non-obese participants and 2000 mg daily for obese participants, starting from the second week of pregnancy until delivery. The goal is to evaluate the effectiveness of Glucophage in improving pregnancy outcomes for women with PCOS, including reducing early pregnancy loss, preterm delivery, gestational diabetes, and intrauterine growth restriction.
  Interventions: Procedure: Metformin (Glucophage)
- Standard Care Group: (Active Comparator): Participants in this arm will receive a standard diet and exercise plan but will not receive any pharmacological intervention. This group will serve as a comparison to assess the impact of Glucophage on pregnancy outcomes in women with PCOS. All participants will be closely monitored throughout the pregnancy with regular follow-up visits and ultrasounds.
  Interventions: Procedure: Standard Care (Diet and Exercise Only)

INTERVENTIONS:
Procedure: Metformin (Glucophage) — In this intervention, participants will receive oral metformin (500 mg daily, gradually increasing to 1500 mg daily for non-obese participants and 2000 mg daily for obese participants) starting from the second week of pregnancy and continuing until delivery. Metformin will be administered in combination with a standard diet and exercise plan. The intervention aims to evaluate the impact of metformin on pregnancy outcomes in women with polycystic ovarian syndrome (PCOS), focusing on reducing complications such as early pregnancy loss, preterm delivery, gestational diabetes, and intrauterine growth restriction. Participants will be regularly monitored with follow-up visits, ultrasounds, and glucose tests to assess the effectiveness of the treatment.
  Arms: Glucophage Treatment Group
Procedure: Standard Care (Diet and Exercise Only) — In this intervention, participants will receive a standard diet and exercise plan designed to promote a healthy pregnancy. This intervention does not include any pharmacological treatment, such as metformin. The goal is to evaluate the pregnancy outcomes in women with polycystic ovarian syndrome (PCOS) managed with lifestyle modifications alone, without the added effect of medication. Participants will be monitored through regular follow-up visits, ultrasounds, and glucose tests to track pregnancy progress, including the occurrence of gestational diabetes, preterm delivery, early pregnancy loss, and fetal growth restriction.
  Arms: Standard Care Group:

SUMMARY:
The goal of this clinical trial is to learn if Glucophage (metformin) improves pregnancy outcomes in women with polycystic ovarian syndrome (PCOS). It will also evaluate the safety of Glucophage during pregnancy. The main questions it aims to answer are:

Does Glucophage reduce the risks of early pregnancy loss, preterm delivery, and gestational diabetes? Are there any medical problems associated with taking Glucophage during pregnancy? Researchers will compare Glucophage with standard care (diet and exercise) to see if it improves pregnancy outcomes in women with PCOS.

Participants will:

Take Glucophage or follow a standard diet and exercise plan throughout pregnancy.

Attend regular follow-up visits for checkups, ultrasounds, and blood tests. Have their pregnancy outcomes, such as fetal growth and gestational diabetes, recorded.

DETAILED DESCRIPTION:
This randomized controlled trial aims to evaluate the effectiveness of Glucophage (metformin) in improving pregnancy outcomes for women with polycystic ovarian syndrome (PCOS). The study compares two groups: one receiving standard diet and exercise along with Glucophage and another receiving only standard diet and exercise. Outcomes such as early pregnancy loss, preterm delivery, gestational diabetes, intrauterine growth restriction, and fetal malformations will be assessed.

Participants will be enrolled during their first trimester and followed through delivery. Data will be collected during regular follow-up visits, including ultrasound scans and oral glucose tolerance tests. The study will use statistical analysis to determine whether Glucophage significantly improves maternal and fetal health outcomes compared to standard care. Findings will help guide clinical management strategies for PCOS during pregnancy.

ELIGIBILITY:
Inclusion Criteria:

Pregnant females aged 18-40 years Diagnosed with polycystic ovarian syndrome (PCOS) before conception, as per operational definition.

Present in the 1st trimester at the booking visit. Singleton fetus on booking scan between 5th to 13th week of gestation.

Exclusion Criteria:

Females who do not give informed consent for follow-up. Females with preeclampsia (BP ≥140/90 mmHg with proteinuria >+1 on dipstick method).

Females already diagnosed with gestational diabetes (OGTT >186 mg/dl). Females already taking trial treatment (as per medical record). Twin pregnancy or abnormal placenta (assessed on ultrasound). Diagnosed hypertensives and diabetic patients.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2025-02-02 (Estimated); Primary Completion 2025-05-25 (Estimated); Study Completion 2025-05-26 (Estimated)

PRIMARY OUTCOMES:
Rate of early pregnancy loss | From enrollment to 24 weeks of gestation.
  The primary outcome of this study is to evaluate the rate of early pregnancy loss in pregnant women with polycystic ovarian syndrome (PCOS) who receive either Glucophage (metformin) or standard care (diet and exercise). Early pregnancy loss is defined as fetal death occurring before 24 weeks of gestation.

IPD SHARING:
Plan to Share IPD: Undecided